CLINICAL TRIAL: NCT00587574
Title: Prospective Phase II Study for Assessment of Regulatory Immune Cell Populations After Allogeneic Hematopoietic Stem Cell Transplantation and Immunomodulatory Consequences of Chronic Graft-Versus-Host Disease and Therapy
Brief Title: Prospective Phase II Study for Assessment of Regulatory Immune Cell Populations After Allogeneic HSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Christoph Zielinski, Professor, Medical University of Vienna
Other Study IDs: 488/2007; EK Nr 488/2007
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-10

CONDITIONS: Allogeneic Hematopoietic Cell Transplant Recipients
Keywords: chronic graft-versus-host disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells as cell pellets and DNA, plasma and serum samples, tissue biopsy samples, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- I: Chronic graft-versus-host disease
- II: No chronic graft-versus-host disease

SUMMARY:
Allogeneic hematopoietic cell transplantation offers high cure rates for patients with hematological and oncological diseases. Graft-versus-host disease (attack of donor's white blood cells on patient's tissues) is a serious complication also affecting the patient's immune system. Therefore, patients in the early phase after allogeneic cell transplantation are at high risk for severe infectious complications. So far, no predictive biomarkers for the development of the chronic form of graft-versus-host disease are available. By analysing serially immune cell populations of the peripheral blood we will investigate whether certain subsets of cells are associated with development of chronic graft-versus-host disease. In addition, the patients' immune regeneration will be evaluated by serial analyses of peripheral blood immune cell populations 3 months to 2 years after allogeneic cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Receiving grafts from either HLA-identical sibling donors or HLA-matched unrelated donors
* Receiving grafts from HLA-mismatched sibling donors or HLA-mismatched unrelated donors
* Receiving either bone marrow, peripheral blood stem cells or cord blood grafts
* Alive on day 100 after transplant
* Age 18 years or above
* Signed written informed consent

Exclusion Criteria:

* Lymphocytopenia not allowing immunophenotyping
* Treatment with rituximab after HSCT until study entry
* Hepatitis B and C, HIV infection
* Secondary posttransplant malignancies including EBV-lymphoproliferative disease
* Karnofsky score of 30 or below
* Absence of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients after allogeneic hematopoietic cell transplantation
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of perturbed B cell homeostasis with chronic graft-versus-host disease activity of immune system | October 2007 until December 2010

SECONDARY OUTCOMES:
Difference of time-dependent pattern of immune reconstitution after allogeneic cell transplantation between patients with and without chronic graft-versus-host disease | October 2010 until December 2010
Compare number of clinically defined bacterial, viral and fungal infectious episodes between patients with and without chronic graft-versus-host disease | October 2007 until December 2010
Compare the number of circulating T, DC, NK subsets in patients with and without chronic GVHD to identify their respective role in development and prolongation of chronic GVHD | October 2007 until December 2010
Investigate the impact of different immunosuppressive/immunomodulatory treatments for chronic GVHD on various immune cell populations | October 2007 until December 2010
Assess the chimerism of antigen-presenting cells in circulation and tissue specimens and correlate it with occurrence of chronic GVHD | October 2007 until December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Hildegard T Greinix, Professor, Principal Investigator — Medical University of Vienna
Locations (2):
- Medical University of Vienna, Vienna, Austria
- Institute of Hematology and Blood Transfusions Prague, Prague, Czechia